CLINICAL TRIAL: NCT06730633
Title: Implementation of Heart Matters Evidence-based Program
Brief Title: Collaborate and Leverage Evidence in African American Rural Network
Acronym: Co-LEARN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Project Momentum, Inc. (Industry); James McFarlin Community Development, Inc. (Other); Opportunities Industrialization Center, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-1366; 5R01HL157255 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
Keywords: Heart health; Behavioral modification; Community-based participatory research
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Permadyne Premier

STUDY DESIGN:
Intervention Model Description: Non-randomized, propensity-matched-controlled trial. Specifically, 70 participants from the present study will be propensity-matched with 70 participants from NCT02707432.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive the Heart Matters intervention, delivered by community-based facilitators. All participants consenting to the present study will be assigned to this arm.
  Interventions: Behavioral: Heart Matters
- Propensity-matched Control Group (Retrospective) (Active Comparator): This group received the Heart Matters intervention, delivered by researchers, under NCT02707432.
  Interventions: Behavioral: Heart Matters

INTERVENTIONS:
Behavioral: Heart Matters — Heart Matters is a lifestyle modification intervention guided by the theory of planned behavior. Designed to mitigate cardiovascular disease risk factors, the program strives to help participants consume nutritious foods, engage in a more active lifestyle, lose weight and lower their systolic or diastolic blood pressure. Lifestyle modifications can include weight loss, a reduction in percent calorie fat consumption and total sodium intake, improving diet and increasing physical activity, and reducing daily alcoholic beverage consumption.
  Other Names: PREMIER

SUMMARY:
The goal of this non-randomized, propensity-matched-controlled study is to assess the effectiveness of the Heart Matters evidence-based program -- previously evaluated for feasibility and efficacy in NCT02707432 -- in improving cardiovascular health outcomes (change in systolic and diastolic blood pressure, primary outcomes) when implemented by community-based facilitators.

DETAILED DESCRIPTION:
The research team will use a non-randomized, propensity-matched-controlled design to evaluate the effectiveness of the Heart Matters evidence-based program -- previously evaluated for feasibility and efficacy under NCT02707432 -- in improving cardiovascular health outcomes when scaled in multiple rural, eastern North Carolina counties and implemented by community-based facilitators.

This study aims to recruit 210 participants, 70 of whom will be propensity-score-matched with participants from NCT02707432. Propensity-score-matching will allow for flexibility in recruitment, statistical rigor, and resource efficiency. The research team hypothesizes that matched participants in the present study will show significant improvements in health outcomes (systolic blood pressure, diastolic blood pressure) compared to the matched NCT02707432 controls.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black or African American
* Reside in rural, eastern North Carolina
* Self-report at least one cardiovascular disease risk factor, such as pre-diabetes, pre-hypertension or stage one hypertension, obesity, or family history of early heart disease

Exclusion Criteria:

* Evidence of active or unstable cardiovascular disease
* Cognitive impairment that limits informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2025-02-22 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean change from Baseline, Systolic Blood Pressure | Baseline, 6 Months
  Blood pressure is measured as the average of three readings, taken in a seated position using an Omron BP6100 digital blood pressure monitor. Reporting will compare participants in the present study with propensity-score-matched controls.
Mean change from Baseline, Diastolic Blood Pressure | Baseline, 6 Months
  Blood pressure is measured as the average of three readings, taken in a seated position using an Omron BP6100 digital blood pressure monitor. Reporting will compare participants in the present study with propensity-score-matched controls.

SECONDARY OUTCOMES:
Number of Participants with Personal History of Cardiovascular Disease | Baseline
  Personal history of cardiovascular disease is measured via self-report at baseline using an adapted item from My Personal Health Record (MyPHR). Personal history of cardiovascular disease is defined as history of diabetes, heart surgery, high blood cholesterol, high blood pressure, pain or pressure in chest, palpitations, stroke, or other heart condition (including heart attack).
Number of Participants with Family History of Cardiovascular Disease | Baseline
  Family history of cardiovascular disease is measured via self-report using an adapted item from the Women's Health Initiative. Family history of cardiovascular disease is defined as having a parent, full-blooded sibling, or child who has ever had a heart condition, such as heart attack, high blood pressure, or stroke.
Mean Systolic Blood Pressure in mmHg | Baseline, 6 Months, 12 Months
  Blood pressure is measured as the average of three readings, taken in a seated position using an Omron BP6100 digital blood pressure monitor.
Mean Diastolic Blood Pressure in mmHg | Baseline, 6 Months, 12 Months
  Blood pressure is measured as the average of three readings, taken in a seated position using an Omron BP6100 digital blood pressure monitor.
Mean Body-mass Index | Baseline, 6 Months, 12 Months
  Body-mass index (BMI) will be calculated as weight (pounds) * 703 / height^2 (inches).
Mean Weight in Pounds | Baseline, 6 Months, 12 Months
  Weight will be measured via a digital scale.
Mean Waist Circumference in Centimeters | Baseline, 6 Months, 12 Months
  Waist circumference will be measured using inelastic tape.
Mean Total Cholesterol in mg/dL | Baseline, 6 Months, 12 Months
  Total cholesterol is measured via blood sample using a Cholestech LDX analyzer.
Mean High-density Lipoprotein (HDL) Cholesterol in mg/dL | Baseline, 6 Months, 12 Months
  HDL cholesterol is measured via blood sample using a Cholestech LDX analyzer.
Mean Low-density Lipoprotein (LDL) Cholesterol in mg/dL | Baseline, 6 Months, 12 Months
  LDL cholesterol is measured via blood sample using a Cholestech LDX analyzer.
Mean Blood Triglycerides in mg/dL | Baseline, 6 Months, 12 Months
  Blood triglycerides are measured via blood sample using a Cholestech LDX analyzer.
Mean Glycated Hemoglobin (A1C) Score | Baseline, 6 Months, 12 Months
  A1C is measured via blood sample using A1CNow+ test kits.
Number of Participants by Categorical Smoking Status | Baseline, 6 Months, 12 Months
  Smoking status is measured via self-report using excerpted items from wave 1 of the Population Assessment of Tobacco and Health Study. Reporting will include number of participants endorsing ever having smoked a cigarette and (among participants who have endorse ever having smoked) numbers of participants endorsing now smoking every day, some days, or not at all.
Mean Healthy Days | Baseline, 6 Months, 12 Months
  Healthy Days measured via self report using the Center for Disease Control (CDC)'s 4-item Healthy Days Core Module (HRQOL-4) with a look-back period of 30 days. HRQOL-4 scores can range from 0 to 30, with 30 indicating maximum number of healthy days.
Mean Heart Disease Fact Questionnaire Score | Baseline, 6 Months, 12 Months
  Heart disease knowledge is measured via self-report using the 25-item Heart Disease Fact Questionnaire (HDFQ). HDFQ scores can range from 0 to 25, with higher scores indicating greater knowledge of heart disease.
Mean University of Rhode Island Change Assessment Score | Baseline, 6 Months, 12 Months
  Readiness for behavioral change is measured via self-report using the 32-item University of Rhode Island Change Assessment (URICA). URICA scores can range from -2 to +14, with higher scores indicating greater levels of readiness to change.
Mean Perceived Stress Scale Score | Baseline, 6 Months, 12 Months
  Perceived stress is measured via self-report using the 10-item Perceived Stress Scale (PSS). PSS scores can range from 0 to 40, with higher scores indicating higher levels of perceived stress.
Mean Alcohol Use Disorders Identification Test - Consumption (AUDIT-C) Score | Baseline, 6 Months, 12 Months
  Alcohol use is measured via self-report using the 3-item Alcohol Use Disorders Identification Test - Consumption (AUDIT-C). AUDIT-C scores can range from 0 to 12, with higher scores indicating greater of drinking quantity and/or frequency.
Mean Minutes of Light, Moderate, and Vigorous Leisure-Time Physical Activity | Baseline, 6 Months, 12 Months
  Minutes of light, moderate, and vigorous leisure-time physical activity is measured via self-report using an English-language version of Registre Gironí del Cor (REGICOR) with a look-back period of one month.
Number of Participants by Categorical Frequency of Dietary Intake of Sweetened Fruit Drinks | Baseline, 6 Months, 12 Months
  Dietary intake of sweetened fruit drinks is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of 100% Pure Fruit Juice | Baseline, 6 Months, 12 Months
  Dietary intake of 100% pure fruit juice is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Soda | Baseline, 6 Months, 12 Months
  Dietary intake of soda is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Water | Baseline, 6 Months, 12 Months
  Dietary intake of water is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Fruit | Baseline, 6 Months, 12 Months
  Dietary intake of fruit is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Vegetables (Excluding Potatoes) | Baseline, 6 Months, 12 Months
  Dietary intake of vegetables (excluding potatoes) is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Frozen and Fast Food | Baseline, 6 Months, 12 Months
  Dietary intake of frozen and fast food is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Processed Meat | Baseline, 6 Months, 12 Months
  Dietary intake of processed meat is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Whole Grains | Baseline, 6 Months, 12 Months
  Dietary intake of whole grains is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Candy, Desserts, and Chocolate | Baseline, 6 Months, 12 Months
  Dietary intake of candy, desserts, and chocolate is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Chips | Baseline, 6 Months, 12 Months
  Dietary intake of chips is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Sugary Cereals | Baseline, 6 Months, 12 Months
  Dietary intake of sugary cereals is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Fish | Baseline, 6 Months, 12 Months
  Dietary intake of fish is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Nuts and Seeds | Baseline, 6 Months, 12 Months
  Dietary intake of nuts and seeds is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.
Number of Participants by Categorical Frequency of Dietary Intake of Eggs | Baseline, 6 Months, 12 Months
  Dietary intake of eggs is measured via an adapted self-report item from Family Life, Activity, Sun, Health, and Eating (FLASHE) with a look-back period of 7 days. Reporting will include categorical number of participants endorsing non-consumption, 1-3 times weekly consumption, 4-6 times weekly consumption, once-daily consumption, twice-daily consumption, or three-or-more times daily consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Dave, MBBS, DrPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (9):
- United States (9):
  - A Better Chance, A Better Community, Enfield, North Carolina
  - The Mercer Foundation, Inc., Nashville, North Carolina
  - Marks Chapel Baptist Church, Rocky Mount, North Carolina
  - Thorne's Chapel Missionary Baptist Church, Rocky Mount, North Carolina
  - Truth Tabernacle Ministries, Rocky Mount, North Carolina
  - Girls Making the Grade, Rocky Mount, North Carolina
  - Carolina Hierarchy of Needs, Spring Hope, North Carolina
  - St. James United Holy Church, Stantonsburg, North Carolina
  - Warren County Health Department, Warrenton, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with The University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with The University of North Carolina at Chapel Hill

DOCUMENTS (1):
  • Informed Consent Form (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT06730633/ICF_000.pdf